CLINICAL TRIAL: NCT00254709
Title: Open, Pilot, Comparative Study to Evaluate the Efficacy and Safety of Two Immunosuppressor Regimens, Anti Il-2, Sirolimus Mycophenolate, Mophetyl and Steroids Versus Sirolimus, Cyclosporine, and Withdrawal of Cyclosporine Since the Third Month and Steroids in Elderly Population
Brief Title: Study Evaluating Two Different Sirolimus-based Immunosuppressive Regimens in Elderly Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0468-100970
Record Dates: First submitted 2005-11-11; First posted 2005-11-16 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Kidney Failure; Graft Rejection; Aged
Keywords: kidney transplant; elderly
MeSH Terms: conditions — Renal Insufficiency | interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
The purpose of this study is to test two different sirolimus-based immunosuppressive regimens for elderly kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease
* Kidney transplantation
* Both donor and recipient older than 60 years

Exclusion Criteria:

* Prior or concurrent transplant of any organ other than the kidney
* Current clinically significant infections

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-10; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Renal function at 3 and 12 months; measured by Cockroft-Gault formula or serum creatinine

SECONDARY OUTCOMES:
Incidence of acute rejections at 3 and 12 months
Patient and graft survival at 3 and 12 months
Incidence and duration of episodes of acute tubular necrosis
Time to recover renal function (creatinine< 2 mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer